CLINICAL TRIAL: NCT00801333
Title: Derivation of Induced Pluripotent Stem Cells From an Existing Collection of Human Somatic Cells
Status: Recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Benjamin Reubinoff, Professor, Hadassah Medical Organization
Other Study IDs: 0511-08-HMO
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Existing banks of collected cells maintained.

SUMMARY:
Induced pluripotent stem cells potentially may be useful in the future as an unlimited source of cells for transplantation.

The major goal of the project is to develop human iPS cells from various types of cell cultures or lines from existing collections. The IPS cells will be developed for modeling diseases, for developing the technology that may eventually allow the use of IPS cells for transplantation therapy, and for basic research.

DETAILED DESCRIPTION:
The potential to reprogram somatic cells into an embryonic state raises multiple basic research questions related both to the process of reprogramming and the properties of iPS cells. We will use various approaches to study the molecular mechanisms and processes that occur during reprogramming. We will use various experimental systems to characterize and study the properties of the iPS cells, their biology, developmental potential, capability to give rise to functional differentiated progeny etc.

We will induce the differentiation of the iPS cells towards specific cell lineages and the progeny can be used to study the pathogenesis of diseases. They will be used for developing new therapeutic approaches and for high throughput screening of factors for potential toxic or therapeutic effects.

All samples will be non-identified.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers
* Male and Female

Exclusion Criteria:

* Below the official age of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will use human somatic cells from existing collections.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2008-11 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin E Reubinoff, MD PhD, Principal Investigator — Chairman of Department of Obstetrics & Gynecology/IVF, Hadassah Ein Kerem
Locations (2):
- Israel (2):
  - Hadassah Medical Organization - Ein Kerem Campus, Jerusalem
  - Hadassah Ein Kerem, Jerusalem

REFERENCES:
- [Background] Dimos JT, Rodolfa KT, Niakan KK, Weisenthal LM, Mitsumoto H, Chung W, Croft GF, Saphier G, Leibel R, Goland R, Wichterle H, Henderson CE, Eggan K. Induced pluripotent stem cells generated from patients with ALS can be differentiated into motor neurons. Science. 2008 Aug 29;321(5893):1218-21. doi: 10.1126/science.1158799. Epub 2008 Jul 31. PMID 18669821